CLINICAL TRIAL: NCT02877238
Title: Protection by Remote Ischemic Preconditioning During Congenital Cardiac Defects Repair Surgery With Sevoflurane But Not Propofol -A Clinical Trial
Brief Title: Remote Preconditioning and Myocardial Protection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sayed Kaoud Abd-Elshafy, Associate profossor of anesthesia, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IIRB0000871234
Record Dates: First submitted 2016-08-15; First posted 2016-08-24 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Congenital Heart Disease
Keywords: remote ischemic preconditioning; sevoflurane; total intravenous anesthetic
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Sevoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): Sevoflurane plus remote ischemic preconditioning anesthesia will be induced and maintain with sevoflurane in addition to remote ischemic preconditioning which will be done after induction and before cardiopulmonary bypass by inflating the cuff of blood pressure above 200mmhg in the lower limb every 5 min for 3 cycles
  Interventions: Drug: Sevoflurane plus remote ischemic preconditioning
- Group B (Active Comparator): anesthesia will be induced and maintain with total intravenous anesthesia (propofol, midazolam plus fentanyl) during plus remote ischemic preconditioning in addition to remote ischemic preconditioning which will be done after induction and before cardiopulmonary bypass by inflating the cuff of blood pressure above 200mmhg in the lower limb every 5 min for 3 cycles
  Interventions: Drug: Total intravenous anesthesia plus remote ischemic preconditioning

INTERVENTIONS:
Drug: Sevoflurane plus remote ischemic preconditioning — Inhalational anesthesia (Sevoflurane) in addition to remote ischemic preconditioning
  Other Names: Group A
  Arms: Group A
Drug: Total intravenous anesthesia plus remote ischemic preconditioning — Total intravenous anesthesia (propofol plus fentanyl) in addition to remote ischemic preconditioning
  Other Names: Group B
  Arms: Group B

SUMMARY:
Remote ischemic preconditioning (RIPC) of the myocardium by limb ischemia/reperfusion may mitigate cardiac damage, but its interaction with the anesthetic regimen is unknown.

DETAILED DESCRIPTION:
The investigators will test if RIPC will be associated with differential effects depending on background anesthesia. Specifically, the investigators hypothesized that RIPC during sevoflurane anesthesia attenuates myocardial injury in patients undergoing congenital cardiac defects repair surgery and that effects may be different during propofol anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric scheduled for cardiac surgery requiring the cardioplegic arrest and cardiopulmonary bypass

Exclusion Criteria:

* Previous cardiac surgery
* Urgent or emergent cases
* Patient with the following diseases diabetes mellitus ,hypertension ,renal failure, hepatic and pulmonary diseases

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2016-08; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Troponin I levels | within first 24 hours after cardiac surgery
  The investigators will obtain blood samples for troponin I level pre-Cardiopulmonary bypass, 6, 12 and 24 hours after the surgery. Troponin I levels, as a marker of myocardial ischemia, have been used in previous adult and pediatric studies on preconditioning.

SECONDARY OUTCOMES:
Highest inotropic score during the first 24 hours after cardiac surgery | within first 24 hours after cardiac surgery
  Inotrope score is a useful predictor of morbidity and mortality in children who undergo heart surgery.
  The inotropic score is calculated as follows: 1 point is assigned for each mcg/kg/min of dopamine and dobutamine, and 10 points is assigned for each 0.1 mcg/kg/min of epinephrine, norepinephrine, and phenylephrine. Inotrope score is a useful predictor of morbidity and mortality in children who undergo heart surgery
Mortality at 30 days | 30 days
  Proportion of patients who dies within 30 days of their surgical repair
Cardiac function | within first 24 hours of cardiac surgery
  Cardiac rhythm on return if it will be sinus rhythm or return with ventricular fibrillation

CONTACTS AND LOCATIONS:
Overall Officials: Sayed K Abd-Elshafy, MD, Principal Investigator — Associate professor of anesthesia
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided